CLINICAL TRIAL: NCT06823258
Title: Pharmacokinetic Study of HS-10365 Capsule in Subjects with Hepatic Impairment and Normal Hepatic Function
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-10365-110
Record Dates: First submitted 2024-12-23; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: NSCLC (advanced Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: HS-10365 160mg (Experimental): Participants with Hepatic Impairment will receive HS-10365 160mg administered orally
  Interventions: Drug: HS-10365
- Arm B: HS-10365 160mg (Experimental): Participants with normal hepatic function will receive HS-10365 160mg administered orally
  Interventions: Drug: HS-10365

INTERVENTIONS:
Drug: HS-10365 — HS-10365 administered orally once at D1

SUMMARY:
This study will be conducted in subjects with moderate Hepatic Impairment, mild hepatic Impairment and normal hepatic function. The study will be conducted in two stages. Based on the research results of moderate hepatic Impairment and matched control subjects with normal hepatic function, the sponsor will make a comprehensive analysis to decide whether it is necessary to conduct a study on the mild hepatic Impairment and matched control subjects with normal hepatic function

ELIGIBILITY:
Inclusion Criteria:

* All participants must meet all of the following conditions:

  1. Voluntarily sign an informed consent form before the start of activities related to this study, understand the procedures and methods of this study, and be willing to strictly follow the clinical study protocol to complete this study;
  2. The subjects agree to have no plans to conceive or donate sperm/eggs within 6 months from the signing of the informed consent form until the last administration, and voluntarily adopt effective contraceptive measures (non-pharmacological contraceptive measures were taken during the study period, as detailed in Appendix 1);
  3. On the day of signing the informed consent form, both males and females must be at least 18 years old;
  4. The weight of male subjects shall not be less than 50 kg, and the weight of female subjects shall not be less than 45 kg; Body mass index (BMI) 18-33 kg/m2 (including both ends);
  5. Creatinine clearance rate (calculated using the Cockcroft Gault formula, see Appendix 2) ≥ 60 mL/min.

Subjects with normal hepatic function must also meet all of the following conditions:

1) When screening, the following demographic matching criteria must be met:

1. BMI matching with the matched hepatic impairment group, with a mean within ± 15% range;
2. Age matching with the matched hepatic impairment group, with a mean of ± 5 years;
3. Gender matching with the matched hepatic impairment group，with the same number of individuals for each gender;

Subjects with liver dysfunction must also meet all of the following conditions:

1. Chronic liver injury caused by primary liver disease (such as hepatitis B, hepatitis C, autoimmune hepatitis, alcoholic liver disease, etc.) in subjects with hepatic impairment classified as A or B by Child Pugh grading (see Appendix 3 for Child Pugh grading).
2. Researchers determine that the hepatic function status of the subjects has been stable for at least 2 months based on their clinical symptoms and other examination results available during screening (as determined by the researchers).
3. Individuals who have a stable medication regimen for treating hepatic impairment, complications, and other accompanying diseases for at least 14 days prior to taking the investigational drug, and whose medication does not require adjustment (including medication type, dosage, or frequency, except for diuretics, insulin, and other medications); Or those who have not taken medication.

Exclusion Criteria:

* All participants who meet the following exclusion criteria are not eligible for this study:

  1. During the screening period, 12 lead electrocardiogram results showed QT interval prolongation (male QTcF>470 ms; female QTcF>480 ms);
  2. Individuals at increased risk of QT interval prolongation (such as heart failure, congenital long QT syndrome, family history of long QT syndrome, refractory hypokalemia, or unexplained sudden death in immediate family members under 40 years old);
  3. Individuals who have previously suffered from cardiovascular diseases (such as organic heart disease, myocardial infarction, angina pectoris, arrhythmia, etc.) and are deemed unsuitable for inclusion by the researchers;
  4. Severe or poorly controlled hypertension, including a history of hypertensive crisis or hypertensive encephalopathy; Within 2 weeks prior to the first administration, adjustments were made to antihypertensive medication due to poor blood pressure control; During the screening period, systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg;
  5. Those who have difficulty swallowing or have undergone surgery that may affect drug absorption, distribution, metabolism, and excretion, and are deemed unsuitable for inclusion by the researchers;
  6. Individuals who are prone to allergic reactions or have an allergic constitution (such as those who are allergic to pollen, two or more drugs/foods), or those who are known to be allergic to the study drug or any component of the study drug;
  7. Individuals who have participated in any other clinical trials within the previous 3 months and have used study drugs or plan to participate in other clinical trials during the study period (those who have not been given the study drug or placebo after enrollment may be included);
  8. Individuals who have donated blood or lost blood ≥ 400 mL within the first 3 months of screening, or have received blood transfusions or used blood products, or intend to donate blood during the trial period or within 1 month after the trial ends;
  9. Individuals who have used strong or moderate inducers or inhibitors of P-gp and/or CYP3A4 enzymes and/or P-gp, BCRP, MATE1 or MATE2-K substrates within the previous month of screening (see Appendix 4);
  10. Prior to administration, any proton pump inhibitors (PPIs), H2 receptor antagonists, local antacids, oral alkaline drugs, or other drugs that reduce gastric acid secretion were used, and HS-10365 was administered within 7 half lives of the aforementioned drugs;
  11. Individuals who have consumed a special diet (including dragon fruit, mango, grapefruit, and/or xanthine diet, chocolate) and/or consumed excessive amounts of tea, coffee, grapefruit/grapefruit juice, and/or caffeinated beverages (an average of 8 or more cups per day, 200 mL per cup) within 2 weeks prior to administration;
  12. Individuals who consume grapefruit or grapefruit products within 48 hours prior to taking the investigational drug;
  13. Screening for alcoholics within the first 3 months, i.e. those who consume more than 14 units of alcohol per week (1 unit=360 mL of beer, 45 mL of strong liquor with an alcohol content of 40%, or 150 mL of wine) or have a positive alcohol screening result;
  14. Individuals who smoke an average of 10 or more cigarettes per day within the first 3 months of screening, or who cannot stop using any tobacco products during the trial period;
  15. Individuals with a history of drug use, substance abuse, or a positive urine drug test;
  16. Individuals who have used vaccines or plan to use vaccines during the study period within 14 days prior to taking the investigational drug;
  17. Pregnant or lactating women, or women of childbearing age who test positive for pregnancy;
  18. Difficulty in venous blood collection and/or unsuitability for receiving venipuncture / indwelling needles;
  19. Due to other reasons, this study may not be completed or the researcher may determine that the participant is not suitable.

Subjects with normal hepatic function should be excluded if they meet any of the following exclusion criteria:

1. History of liver injury;
2. Individuals who have previously or currently suffered from any clinically serious diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry, and metabolic abnormalities, or any other diseases that can interfere with the test results;
3. Abnormalities in physical examination, vital signs, laboratory tests, 12 lead electrocardiogram, chest X-ray, abdominal ultrasound, and other examinations have clinical significance as determined by the researchers;
4. Those who are positive in any index screening of hepatitis B surface antigen, hepatitis C antibody, HIV antigen/antibody or Treponema pallidum antibody;
5. Individuals who have used any prescription drugs, over-the-counter drugs, herbal medicines, or health supplements (excluding topical preparations that exert local effects) within 14 days prior to drug administration.

If a subject with hepatic impairment meets any of the following exclusion criteria, they should be excluded:

1. The subject has any of the following conditions: ① Having undergone liver transplantation in the past; ② Having undergone partial hepatectomy in the past; ③ Patients who are suspected of or diagnosed with liver cancer or other malignant tumors (except for specific cancers that have been surgically removed and completely cured, such as basal cell carcinoma or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix; except for patients with liver cancer who have received radical treatment and have no recurrence; except for patients with liver cancer at BCLC stage 0)；④ Patients with liver failure; ⑤ Those who had rupture and bleeding of esophageal and gastric varices within 3 months before screening; ⑥ Patients with biliary cirrhosis, extrahepatic biliary obstruction and other diseases, and who are deemed by the investigator as not suitable to participate in this trial;
2. The laboratory test results during screening meet any of the following criteria: (a) alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>10 × ULN; (b) Absolute neutrophil count (NE #)<0.75 × 109/L; (c) Hemoglobin (HGB)<60 g/L; (d) Alpha fetoprotein (AFP)>100 ng/mL;
3. Individuals who test positive for HIV antigen/antibody screening; If the Treponema pallidum antibody is positive, the Rapid Plasma Reactive Protein (RPR) test should be added. If RPR is also positive, it should be excluded;
4. In addition to the primary liver disease itself, those who have previously or currently suffered from other serious organ systemic diseases, including but not limited to uncontrollable gastrointestinal, respiratory, renal, neurological, blood, endocrine, tumor, immune, psychiatric or cardiovascular diseases, or clinical laboratory tests that have clinical significance and have been determined by the research doctor to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of HS-10365 | From the first dose (Day 0) up to Day 6
Pharmacokinetic parameters AUC0-t of HS-10365 | From the first dose (Day 0) up to Day 6
Pharmacokinetic parameters AUC0-∞ of HS-10365 | From the first dose (Day 0) up to Day 6

SECONDARY OUTCOMES:
Safety : the Incidence rate of AE related to Clinical symptoms | From the first dose (Day 0) up to Day 6
Safety：the incidence rate of Laboratory ABNORMALITIES | From the first dose (Day 0) up to Day 6
the incidence rate of adverse events/serious adverse events | From the first dose (Day 0) up to Day 6